CLINICAL TRIAL: NCT00672568
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Two-Stage Exploratory Study to Evaluate Safety, Tolerability, Efficacy, and Pharmacokinetics of Intraoperative Subacromial Injection With 4975 in Patients Undergoing Arthroscopic Rotator Cuff Repair of the Shoulder
Brief Title: Safety and Tolerability of 4975 in Patients Undergoing Arthroscopic Surgery to Repair the Rotator Cuff of the Shoulder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been halted after completing Stage 1, for corporate reasons. No future patients will be enrolled or treated.
Sponsor: Anesiva, Inc. (Industry)
Responsible Party: Shaun Comfort, MD, Anesiva, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114-04P
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Rotator Cuff Repair of the Shoulder
Keywords: Rotator cuff, Shoulder, Arthroscopic shoulder surgery
MeSH Terms: interventions — ALGRX-4975

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 4975
  Interventions: Drug: 4975 - Highly purified capsaicin
- 2 (Experimental): 4975
  Interventions: Drug: 4975 - Highly purified capsaicin
- 3 (Experimental): 4975
  Interventions: Drug: 4975 - Highly purified capsaicin
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4975 - Highly purified capsaicin — Solution, 0.5 mg, single dose, injection
  Other Names: Adlea
  Arms: 1
Drug: 4975 - Highly purified capsaicin — Solution, 0.75 mg, single dose, injection
  Other Names: Adlea
  Arms: 2
Drug: 4975 - Highly purified capsaicin — Solution, 0.1 mg, Single dose, injection
  Other Names: Adlea
  Arms: 3
Drug: Placebo — Solution, single dose, injection
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and explore the efficacy of a single intraoperative injection of 4975 in patients undergoing arthroscopic surgery for rotator cuff repair of the shoulder

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, two-stage exploratory study in patients undergoing arthroscopic rotator cuff repair surgery.

Stage 1) Patients will be randomized to receive either 4975 or placebo. The dose of 4975 will be escalated in a protocolized manner based on safety and tolerability.

Stage 2) Patients will be randomized in a 1:1 ratio to receive either the selected dose of 4975 or placebo. All patients will be observed in the hospital for at least two days following surgery for safety, tolerability, and efficacy assessments. In addition there will be two planned follow-up visits after hospital discharge.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between the ages of 18 and 75 inclusive
* In overall good health and planning to undergo unilateral arthroscopic shoulder surgery to repair at least one rotator cuff tendon involving humeral attachment
* Willing and able to complete the study procedures, pain assessments, and medication diaries, and to communicate in Korean or English with study personnel

Key Exclusion Criteria:

* Shoulder surgery requiring concomitant repair of biceps muscle or associated tendon(s)
* Planning to undergo shoulder surgery on both shoulders
* Use of disallowed pain medications prior to the surgery
* Female patients who are pregnant or lactating or who plan to get pregnant
* Diabetes mellitus with a known HbA1C>9.5

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity using a standard 11-point numerical rating system (NRS), which will be assessed at predefined times following surgery | 28 Days

SECONDARY OUTCOMES:
Mean overall daily pain and worst daily pain. Pain intensity with physical therapy. Safety outcomes include ECG, vital signs, adverse drug reactions, and wound exams | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Comfort, MD, Study Director — Anesiva, Inc.
Locations (4):
- South Korea (4):
  - Kyungpook National university Hospital, Daegu, Jung-gu
  - Seoul National University Hospital, Seoul, Kyunggido
  - Gyeongsang National University Hospital, Jinju, Kyungsangnamdo
  - Kangnam St. Mary's Hospital, Seoul, Seocho-gu

REFERENCES:
- See also: Anesiva Home Page — http://www.anesiva.com/wt/page/pipeline
- See also: ADLEA Product Information — http://www.anesiva.com/wt/page/adlea